CLINICAL TRIAL: NCT01731574
Title: An Open-label, Randomized, Three-period Crossover Trial in Healthy HIV-negative Women to Assess the Drug-drug Interaction Between Dapivirine Vaginal Ring-004 and Miconazole Nitrate
Brief Title: DDI Potential: Dapivirine Vaginal Ring and Miconazole Nitrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 028
Record Dates: First submitted 2012-11-14; First posted 2012-11-22 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV
MeSH Terms: interventions — Dapivirine; Miconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapivirine Ring + Miconazole (Active Comparator): Dapivirine Ring + miconazole
  Interventions: Drug: dapivirine; Drug: miconazole
- Dapivirine Ring (Experimental): Dapivirine Ring
  Interventions: Drug: dapivirine

INTERVENTIONS:
Drug: dapivirine
Drug: miconazole
  Arms: Dapivirine Ring + Miconazole

SUMMARY:
This trial will investigate the potential drug-drug interaction between dapivirine vaginal Ring-004 and vaginally administered miconazole nitrate, and will evaluate the safety of co-administration of the dapivirine vaginal ring and miconazole nitrate in healthy, HIV-negative women.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and ≤ 40 years of age who can give written informed consent
2. Available for all visits and consent to follow all procedures scheduled for the trial
3. Healthy, based on medical history, vital signs, physical examination, urinalysis (dipstick and microscopy (if indicated)), laboratory evaluations for genital infections (bacterial vaginosis, gonorrhoea, chlamydia and trichomonas), and laboratory evaluations for haematology and chemistry
4. HIV-negative as determined by an HIV test at the time of enrolment
5. On a stable form of contraception, defined as:

   * A stable oral contraceptive regimen for at least 2 months prior to enrolment, OR
   * Transdermal contraceptive patch for at least 3 months prior to enrolment, OR
   * Long-acting progestins for at least 6 months prior to enrolment, OR
   * An IUD inserted (with no vaginal or gynaecological complaints associated with its use) at least 3 months prior to enrolment, OR
   * Have undergone surgical sterilisation at least 3 months prior to enrolment, AND willing to use oral contraceptives if necessary to delay menstruation during the vaginal sampling period
6. Upon pelvic examination at the time of enrolment, the cervix and vagina appear normal as determined by the Investigator/Physician
7. Asymptomatic for genital infections at the time of enrolment (if a woman is diagnosed with any treatable STI, either clinically or by laboratory test at the time of screening, she must receive treatment at least 2 weeks prior to enrolment)
8. Willing to refrain from the use of topical medications, vaginal products or objects, including female condoms, tampons, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 14 days prior to enrolment and for the duration of the trial.
9. Documentation of no abnormality on cervical cytology, including grossly bloody smear, within 90 days prior to screening
10. Willing to refrain from participation in any other research trial for the duration of this trial
11. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, e.g. by home visit or telephone, or via family or close neighbour contacts (confidentiality to be maintained)
12. Willing to agree to abstain from all the following for a total of 2 days (48 hours) prior to each trial visit:

    * Penile-vaginal intercourse
    * Oral contact with her genitalia
13. Hepatitis B and C negative at the time of enrolment.

Exclusion Criteria:

1. Currently pregnant or had their last pregnancy outcome within 3 months prior to screening
2. Currently breast-feeding
3. Currently or within two months of participation in any other clinical research trial involving investigational or marketed products prior to screening
4. Untreated symptomatic urogenital infections, e.g. urinary tract or other sexually transmitted infections, or other gynaecological conditions such as vaginal itching, pain, or discharge, within 2 weeks prior to enrolment
5. Have a Grade 2 or higher pelvic examination finding, according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
6. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence
7. Current vulvar or vaginal symptoms/abnormalities that could influence the trial results
8. Cervical cytology at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation
9. Symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection
10. Any Grade 2, 3 or 4 haematology, biochemistry or urinalysis laboratory abnormality at baseline (screening) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
11. Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment
12. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone
13. Any serious acute, chronic or progressive disease (e.g. any known history of neoplasm, cancer, diabetes, epilepsy, cardiac disease, autoimmune disease, HIV, AIDS, or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition
14. Have undergone a hysterectomy
15. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Dapivirine Area under the concentration time curve (AUC) | 24 hr, 14 days, and 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Sciences, Lange Beeldekensstraat 267, Antwerpen, Belgium